CLINICAL TRIAL: NCT06305663
Title: A Multi-center, Randomized, Parallel, Bilateral, Investigator-masked Study to Evaluate the Safety and Efficacy of the Bausch + Lomb Myopia Control Lens for the Correction of Myopic Ametropia and Slowing the Progression of Myopia in Children
Brief Title: A Study to Evaluate the Safety and Efficacy of the Bausch + Lomb Myopia Control Lens for the Correction of Myopic Ametropia and Slowing the Progression of Myopia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 921
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The identity of the study eye will be masked to subjects, assessors, and other masked personnel while masking is maintained..
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bausch + Lomb (kalifilcon A) Myopia Control Soft (Hydrophilic) (Experimental)
  Interventions: Device: Bausch + Lomb (kalifilcon A) Myopia Control Soft (Hydrophilic)
- CooperVision MiSight (omafilcon A/60%) Myopia Control one day Soft Contact Lens (Active Comparator)
  Interventions: Device: CooperVision MiSight (omafilcon A/60%) Myopia Control one day Soft Contact Lens

INTERVENTIONS:
Device: Bausch + Lomb (kalifilcon A) Myopia Control Soft (Hydrophilic) — Bausch + Lomb (kalifilcon A) Myopia Control Soft (Hydrophilic)
  Arms: Bausch + Lomb (kalifilcon A) Myopia Control Soft (Hydrophilic)
Device: CooperVision MiSight (omafilcon A/60%) Myopia Control one day Soft Contact Lens — CooperVision MiSight (omafilcon A/60%) Myopia Control one day Soft Contact Lens
  Arms: CooperVision MiSight (omafilcon A/60%) Myopia Control one day Soft Contact Lens

SUMMARY:
A Study to Evaluate the Safety and Efficacy of the Bausch + Lomb Myopia Control Lens for the Correction of Myopic Ametropia and Slowing the Progression of Myopia in Children

DETAILED DESCRIPTION:
A Multi-center, Randomized, Parallel, Bilateral, Investigator-masked study to Evaluate the Safety and Efficacy of the Bausch + Lomb Myopia Control Lens for the Correction of Myopic Ametropia and Slowing the Progression of Myopia in Children

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 8 to 12 years plus 11 months old on the date the Informed Assent and Parental or Guardian Informed Consent are signed and have capacity to provide voluntary informed consent.
2. Subject must meet the following determined by cycloplegic subjective refraction in both eyes at screening:

   1. Spherical Equivalent Refractive Error (SERE): between -0.75 D and -4.00 D, inclusive.
   2. Astigmatism: ≤ -0.75 D. c. Anisometropia: < 1.00 D.
3. Subject must be myopic and require lens correction from -0.75 D to -4.00 D, at screening, in each eye.
4. Subject must have distance best-spectacle corrected visual acuity (BSCVA) by non-cycloplegic manifest refraction of +0.04 logMAR (20/20 Snellen equivalent) or better in each eye.
5. Subject and Parent or Guardian must be willing to participate in either the test or the comparator assignment.
6. Subject agrees to wear the assigned contact lenses for a minimum of 10 hours per day, at least 6 days per week, for the duration of the 24-month study.
7. Subject must have wearable and visually functioning eyeglasses.
8. Subject must be in good general health according to their and parent's or guardian's knowledge

Exclusion Criteria:

1. Subject has previously worn, or currently wears rigid gas permeable contact lenses, including orthokeratology lenses.
2. Current or prior use of bifocals, progressive addition lenses, multifocal soft contact lenses, atropine, pirenzepine or ANY other myopia control treatment.
3. Subject appears to exhibit poor personal hygiene (that in the Investigator's opinion might prevent safe contact lens wear).
4. Per oral inquiry from parents/guardian, the subject was born earlier than 30 weeks or weighed less than 1,500 g at birth.
5. Prior strabismus, intraocular, or refractive surgery.
6. Subject using any systemic or local eye medication that interfere with the wearing of corneal contact lenses, pupil size, adjustment or refractive status, or require the removal of lenses during the day".
7. A known allergy to fluorescein, benoxinate, proparacaine, or cyclopentolate.
8. A history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, ocular viral or fungal infections or other recurrent ocular infections.
9. Strabismus by cover test at far (4 m) or near (40 cm) wearing distance correction.
10. Known ocular or systemic disease such as, but not limited to: anterior uveitis or iritis, episcleritis or scleritis, glaucoma, Sjögren's syndrome, lupus erythematosus, scleroderma, or diabetes.
11. At the discretion of the Investigator, any ocular, systemic or neuro developmental conditions that could influence refractive development such as, but not limited to: persistent pupillary membrane, vitreous hemorrhage, cataract, corneal scarring, ptosis, eyelid hemangiomas, Marfan's syndrome, Down syndrome, Ehlers-Danlos syndrome, Stickler syndrome, ocular albinism, retinopathy of prematurity. Subjects with trichiasis, that in the Investigator's judgement does not interfere with contact lens wear, are eligible for this study.
12. Keratoconus or an irregular cornea.
13. Subjects with any Grade 2 or greater finding during the slit lamp examination, or subjects with any scar or neovascularization within the central 6 mm of the cornea, or subjects with corneal infiltrates, of ANY GRADE.
14. Subjects with any "present" finding during the slit lamp examination (biomicroscopy) that, in the investigator's judgment, interferes with contact lens wear. Subjects with minor peripheral corneal scarring (that does not extend into the central area), that in the Investigator's judgment does not interfere with contact lens wear, are eligible for this study.
15. The Investigator for any reason considers that it is not in the best interest of the Subject to participate in the study.
16. Subjects participating in any drug clinical investigation within 4 weeks or device clinical investigation within 2 weeks prior to entry into this study (Screening/Dispensing Visit) and/or planning to do so during the period of study participation.
17. Immediate family or close relative is a member of site study team members

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 418 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in axial length. | 1 and 2 years
  Mean change from baseline in axial length will be evaluated at the one-year and two-year visits.
Mean change from baseline in cycloplegic SERE. | 1 and 2 years
  Mean change from baseline in cycloplegic SERE will be evaluated at the one-year and two-year visits.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Site 105, Beijing, Beijing Municipality
  - Site 107, Dongcheng, Beijing Municipality
  - Site 109, Xiamen, Fujian
  - Site 111, Haikou, Hainan
  - Site 110, Wuhan, Hubei
  - Site 102, Shanghai, Shanghai Municipality
  - Site 106, Taiyuan, Shanxi
  - Site 108, Shenzhen, Shenzhen
  - Site 103, Chengdu, Sichaun Province
  - Site 104, Nankai, Tianjin Municipality
  - Site 101, Wenzhou, Zhejiang